CLINICAL TRIAL: NCT03360253
Title: Safety and Efficacy of Lactobacillus Reuteri DSM 17938 to Reduce the Crying Time in Infants With Colic: Randomised Controlled Trial With Two Parallel Arms. Version 3.3. Nov,11th,2016
Brief Title: Clinical Trial of L. Reuteri in Infantile Colic 2017
Acronym: Colic2017
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, MD, MSc, DSc, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Colic2017
Record Dates: First submitted 2017-04-30; First posted 2017-12-04 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind allocation concealment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Children allocated on different arms will receive drops of probiotics or placebo. Both product are identical in appearence and flavor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HMilkProb (Experimental): L. reuteri DSM 17938 in drops will be given at a dose of 5 drops containing 1x108 colony-forming units (CFU) once time per day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together to give the product the correct rheological properties
  Interventions: Dietary Supplement: L. reuteri DSM 17938 in drops
- HMilkPlacebo (Placebo Comparator): The placebo consists of an identical formulation except that the L. reuteri is not present
  Interventions: Other: Placebo
- IFormProb (Experimental): L. reuteri DSM 17938 in drops will be given at a dose of 5 drops containing 1x108 colony-forming units (CFU) once time per day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together to give the product the correct rheological properties
  Interventions: Dietary Supplement: L. reuteri DSM 17938 in drops
- IFormPlacebo (Placebo Comparator): The placebo consists of an identical formulation except that the L. reuteri is not present
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 in drops — L. reuteri DSM 17938 will be given at a dose of 5 drops containing 1x108 colony-forming units (CFU) once time per day in an oil formulation delivered from a drop bottle
  Arms: HMilkProb; IFormProb
Other: Placebo — The placebo consists of an identical formulation except that the L. reuteri is not present
  Arms: HMilkPlacebo; IFormPlacebo

SUMMARY:
RCT to evaluate the safety and efficacy of Lactobacillus reuteri DSM 17938 to significantly reduce the duration of crying time and fussines in infants from 15days to 4 months of age with colic, feed with human milk (30% sample) or infant formula (70%)

DETAILED DESCRIPTION:
RCT to evaluate the safety and efficacy of Lactobacillus reuteri DSM 17938 administrated for 21 days to significantly reduce the duration of crying time and fussines in infants from 15days to 4 months of age with colic. 66 infants feed with human milk and 180 infant feed with infant formula will be included. As primary outcome we will measure the difference between children receiving L. reuteri DSM 17938, 108 CFU vs children receiving placebo regarding average daily crying duration (minutes per day, from average of crying from days 19 to 21 after randomization), measured by Barr diary. Secondary/exploratory outcomes will be average of crying time on day 7 and 14 (Barr diary) of L. reuteri groups vs placebo group; average of crying and fussing time on day 7, 14 and average from days 19 to 21 after randomization (Barr diary) of L. reuteri groups vs placebo group; responders percentage on day 7, 14 and 21, decrease in daily average crying time of 50% during the study; QoL (PedsQL-2.0-Family Impact Module AU2.0 spa-MX) changes from baseline to days 7, 14 and 21 and Edinburg postnatal depression scale for mothers from baseline to days 7, 14 and 21

ELIGIBILITY:
Inclusion Criteria:

* Younger than 10 weeks of age
* Full term infant (37-42 weeks gestational age)
* Birth weight ≥ 2,500g
* Apgar score ≥ 7 at 5 minutes
* Infantile colic diagnosed according to modified Wessel's criteria (crying more than 180 min/day during 3 days for at least a week prior to enrolment)
* Parental motivation to postpone changes in the infant feeding mode, unless necessary
* Stated availability throughout the study period
* Parent(s) willingness and ability to fill out charts and questionnaires
* Signed informed consent

Exclusion Criteria:

* Failure to thrive
* Chronic illness or major medical problem
* Gastrointestinal disease
* Use of any antibiotic 2 weeks before Day 1 in the study. This applies also to lactating mothers whose infants participate in the trial
* Use of supplements/eaten foods that contain Lactobacillus reuteri, 2 weeks before Day 1
* Use of proton pump inhibitors in the week (7 days) prior to enrolment
* If breastfeeding, use of probiotic by the mother in the week (7 days) prior to enrolment and throughout the study period
* Use of infant formula with hydrolysed protein
* Infant receiving solid foods (such as cereals, mashed fruits or vegetable purée)
* Change of feeding mode planned by parents during the study period

Ages: 1 Week to 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Crying time | 21 days
  Difference between children receiving L. reuteri DSM 17938, 108 CFU vs children receiving placebo regarding average daily crying duration (minutes per day, from average of crying from days 19 to 21 after randomization), measured by Barr diary.
  Difference between children receiving L. reuteri DSM 17938, 108 CFU vs children receiving placebo regarding average daily crying duration (minutes per day, from average of crying from days 19 to 21 after randomization), measured by Barr diary.

SECONDARY OUTCOMES:
Preliminary crying time | Day 7 and 14
  Average of crying time on day 7 and 14 (Barr diary) of L. reuteri groups vs placebo group
Crying and fussing | 7,14 and 21 days
  Average of crying and fussing time on day 7, 14 and average from days 19 to 21 after randomization (Barr diary) of L. reuteri groups vs placebo group
Total responders | 7,14 and 21 days
  Responders percentage on day 7, 14 and 21, decrease in daily average crying time of 50% during the study
Impact on Quality of Life | 7, 14 and 21 days
  Impact on Quality of Life measured by PedsQL-2.0-Family Impact Module AU2.0 spa-MX. Changes from baseline to days 7, 14 and 21
Maternal depression | 7, 14 and 21 days
  Maternal depression evaluated with Edinburgh Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez-Castrellon, DSc, Principal Investigator — Hospital General Dr. Manuel Gea Gonzalez
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No